CLINICAL TRIAL: NCT06361082
Title: The Application of Ultrasonic Backscattering Imaging Technique to Patients With Anterior Cruciate Ligament Reconstruction and Shoulder Musculoskeletal Diseases
Brief Title: Ultrasonic Backscatter Imaging for ACL Reconstruction and Shoulder Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CORPG5N0061
Record Dates: First submitted 2024-03-15; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: ACL Injury; ACL Reconstruction
Keywords: Musculoskeletal ultrasound; ultrasound; Back-scattering; ACL reconstruction; ACL injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-ACLR Control Group (No Intervention): Control group arm. Subjects In this arm will receive MRI and ultrasound examination, without receiving any treatment.
- ACLR Intervention Arm (Experimental): Intervention group arm. Subjects In this arm will receive MRI and ultrasound examination, before and after receiving ACL reconstruction.
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — ACL reconstruction
  Arms: ACLR Intervention Arm

SUMMARY:
This study explores ultrasonic scattering imaging technology in patients undergoing anterior cruciate ligament (ACL) reconstruction and those with shoulder musculoskeletal disorders. Ultrasonography, widely utilized for diagnosing musculoskeletal conditions, faces limitations due to factors like operator experience and equipment settings, often lacking in quantifiable disease metrics. Nakagami imaging, employing the backscattering statistical distribution model, offers a quantitative assessment method that minimizes subjective interpretation by extracting tissue properties through the interaction between ultrasound and tissue microstructure. The Nakagami model effectively describes tissue scattering statistics, enabling the identification and classification of tissue features based on specific scattering conditions.

ACL reconstruction is commonly performed, with postoperative complications including joint stiffness and muscle strength decline, associated with changes in muscle quality and volume. Similarly, soft tissue injuries around the shoulder and ankle are prevalent in sports medicine, with ultrasound used to assess the severity of injuries to soft tissues such as the rotator cuff tendons/muscles and surrounding ligaments of the shoulder, as well as the medial and lateral ligament complexes of the ankle. Preliminary findings suggest that Nakagami imaging can differentiate layers within normal tendons, proposing its potential for visualizing and quantifying soft tissue lesions post-ultrasound, aiming for standardized diagnostic criteria.

The results of this project could significantly improve the diagnostic efficacy of musculoskeletal ultrasound, facilitating earlier treatment and reducing the socio-economic impacts. Academically, it positions the investigating team as pioneers in the application of ultrasound inverse scattering imaging technology.

DETAILED DESCRIPTION:
This study aims to explore the application of ultrasonic scattering imaging technology in patients after anterior cruciate ligament (ACL) reconstruction and in patients with shoulder musculoskeletal disorders. Ultrasonography is a convenient, real-time, non-invasive, and portable imaging tool commonly used by clinicians for the diagnosis of musculoskeletal system disorders. However, the interpretation of ultrasound images can be affected by factors such as operator experience, probe orientation, machine type, and parameter settings, and most diseases cannot be quantified. Nakagami imaging, based on the backscattering statistical distribution model, is a quantitative assessment method that can reduce subjective human judgment. It extracts the basic physical properties of tissues based on the interaction between ultrasound and tissue microstructure. The Nakagami distribution is an effective model for describing tissue inverse scattering envelope statistics, which can identify tissue ultrasound image features and classify the examined tissue by comparing it with the specified envelope-related scattering conditions.

ACL reconstruction surgery is a commonly performed procedure. Postoperative issues often include joint stiffness, loss of neuromuscular control, muscle mass loss, and muscle strength decline. Changes in muscle quality and volume are associated with a decrease in thigh muscle strength. Both MRI and ultrasound can be used to assess changes in muscle volume and quality. Soft tissue injuries around the shoulder and ankle joints are common in the field of sports medicine. Ultrasound is commonly used to assess the severity of injuries to soft tissues such as the rotator cuff tendons/muscles and surrounding ligaments of the shoulder, as well as the medial and lateral ligament complexes of the ankle. Preliminary results of this study show that Nakagami scattering imaging can visually distinguish layers within normal tendons. The investigative team hypothesizes that ultrasonic Nakagami scattering imaging can provide a method for visualizing and subsequent quantitative analysis of suspected soft tissue lesions in patients after ultrasound scanning, with the goal of achieving standardized diagnostic parameters for soft tissue lesions.

The results of this project may enhance the diagnostic efficacy of musculoskeletal ultrasound for use in musculoskeletal diseases. If successful, it could lead to earlier diagnosis and treatment for these patients, reducing the socioeconomic losses associated with work and competition. Academically, it would establish the institution and team as world leaders in the application of ultrasound inverse scattering imaging technology.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 and above
* Experimental group: Individuals with tendon, ligament, or nerve disorders around the shoulder joint
* Control group: Individuals with similar age and gender as the experimental group, confirmed by ultrasound and MRI to have no known diseases of the shoulder tendons, ligaments, or nerves

Exclusion Criteria:

* Individuals with a history of injury or disease in the area to be tested: such as fractures, tendon, ligament, or nerve disorders
* Vulnerable groups: such as pregnant women, children, individuals with mental illness, inmates, etc.
* Individuals who cannot communicate in Chinese
* Individuals with poor compliance or obvious mental status abnormalities, or for any reason unable to cooperate with completing clinical symptom interviews, physical examinations, ultrasound examinations, etc.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
MRI of affected limb- Cross sectional area measured in squared cm of quadriceps muscles | 0-6-12 weeks
  MRI of affected limb will be done, to measure quadriceps muscle cross sectional area in with unit of squared centimeters.
Ultrasound Nakagami back scattering analysis- Nakagami index | 0-6-12 weeks
  Ultrasound of affected limb will be done, to calculate Nakagami. A back-scattering analysis algorithm will be applied to derive Nakagami index to give an innovative quantitative assessment of MSK ultrasound. This index as a pure numer index with no unut.

SECONDARY OUTCOMES:
Physical examination of limbs- Angles of Range of Motion of knee | 0-6-12 weeks
  The ROM of knee from affected/control lower limb will be measured with Goniometer and documented in degrees.
MRI of affected limb- Quality of knee structures documented with descriptions for MR signals | 0-6-12 weeks
  MRI of affected limb will be done, to assess muscle quality, and any associate ligamentous change (tendinopathy, tendinosis, etc).
Physical examination of limbs- Laxity of knee ligaments of subjects number with any positive knee physical findings | 0-6-12 weeks
  Any laxity in anterior and posterior cruciate ligaments, medial and lateral collateral ligaments are also be tested and record in (+) or (-) signs.
Ultrasound of affected limb- Cross sectional area measured in squared cm of quadriceps muscles | 0-6-12 weeks
  Ultrasound of affected limb will be done, to measure quadriceps muscle cross sectional area in with unit of squared centimeters.
Ultrasound of affected limb- Quality of knee structures documented with descriptions for echogenicity | 0-6-12 weeks
  Ultrasound of affected limb will be done, to assess muscle quality, and any associate ligamentous change (tendinopathy, tendinosis, etc), in descriptions such as "hypoechoic change, heteroechoic change or eu-echoic appearance"

IPD SHARING:
Plan to Share IPD: No